CLINICAL TRIAL: NCT05485883
Title: A Single-arm Study of the Efficacy of Tislelizumab Combined With Lenvatinib in Patients With Stage III-IV Renal Cancer
Brief Title: Tislelizumab Plus Lenvatinib in Stage III-IV RCC
Acronym: TILUR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILUR
Record Dates: First submitted 2022-07-25; First posted 2022-08-03 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-07

CONDITIONS: Advanced Kidney Cancer
Keywords: Tislelizumab Lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Advanced Renal Cell (Experimental): Patients will receive treatment with Tislelizumab every 3 weeks,and take Lenvatinib 8mg every day
  Interventions: Drug: Tislelizumab Lenvatinib

INTERVENTIONS:
Drug: Tislelizumab Lenvatinib — Patients will receive treatment with Tislelizumab in combination with Lenvatinib every 3 weeks unitl tumor progression or serious side effects

SUMMARY:
This is a phase II study to determine the efficacy and safety of Tislelizumab when given in combination with Lenvatinib as treatment for patients with the advanced kidney cancer . Patients will receive treatment with Tislelizumab in combination with Lenvatinib every 3 weeks unitl tumor progression or serious side effects

DETAILED DESCRIPTION:
This is a phase II study to determine the efficacy and safety of Tislelizumab when given in combination with lenvatinib as treatment for patients with the advanced kidney cancer . Patients will receive treatment with Tislelizumab in combination with lenvatinib every 3 weeks unitl tumor progression or serious side effects.The primary outcome measure was PFS

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Age ≥ 18 years
* Subjects with pathologically and radiologically confirmed renal cell carcinoma: Stage III/IV
* There are no suspected brain metastases
* There are lesions that can be measured by imaging
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Organ function level must meet the following requirements:

Hematological indexes: neutrophil count >= 1.5x10^9/L, platelet count >= 100x10^9/L, hemoglobin >= 9.0 g/dl (can be maintained by blood transfusion); Liver function: total bilirubin <=1.5 ULN, alanine aminotransferase and aspartate aminotransferase <=1.5 ULN

* Women were required to use an effective contraceptive method for three months after the end of the study, and men were required to consent to use an effective contraceptive method with their spouse during and for three months after the end of the study
* The subjects volunteered to join the study, signed informed consent, and had good compliance with follow-up

Exclusion Criteria:

* Prior treatment with radiation, chemotherapy, long-term or high-dose hormone therapy, or immune checkpoint inhibitors
* Previous or concurrent other malignancy
* Previous PD-L1 or PD-L1 treatment, or allergy to PD-L1
* History of primary immunodeficiency
* Active, known or suspected autoimmune diseases
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
* Pregnant or lactating female patients;
* Untreated acute or chronic active hepatitis B or hepatitis C infection. Under the condition of monitoring the virus copy number of patients receiving antiviral treatment, doctors can judge whether they are in line with the patients' individual conditions;
* Have a clear history of active tuberculosis;
* Participating in other clinical researchers;
* Men with reproductive capacity or women who are likely to become pregnant do not take reliable contraceptive measures;
* Uncontrolled concurrent diseases, including but not limited to:

HIV infected (HIV antibody positive); Severe infection in active stage or poorly controlled; Evidence of serious or uncontrollable systemic diseases (such as severe mental, neurological, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension [i.e. hypertension greater than or equal to CTCAE grade 2 after drug treatment]); Patients with active bleeding or new thrombotic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | assessed up to 4 years
  Duration from patient enrollment to disease progression
DCR | assessed up to 4 years
  PerPercentage of evaluable cases in which patients were in remission or stable after treatmen

CONTACTS AND LOCATIONS:
Overall Officials: Changyi Quan, MD,PhD, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Changyi Quan, Tianjin, Tianjin Municipality, China